CLINICAL TRIAL: NCT06786546
Title: Autonomic Control and Vascular Function in Type 1 Diabetes
Brief Title: Type 1 Diabetes Autonomic and Vascular Function
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jasdeep Kaur, Assistant Professor, University of Texas at Austin
Other Study IDs: STUDY00004548
Record Dates: First submitted 2025-01-11; First posted 2025-01-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes (Juvenile Onset); Type 1 Diabetes; Diabetes, Autoimmune
Keywords: autonomic function; exercise pressor reflex; muscle sympathetic nerve activity; Reactive hyperemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for assessing blood glucose, cholesterol, oxidative stress, pro- and anti-inflammatory cytokines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Type 1 Diabetes Group: Men and women diagnosed with Type 1 diabetes
- Healthy Control group: Healthy men and women will be recruited, matched to the Type 1 diabetes group for age, sex and weight

SUMMARY:
The goal of this clinical trial is to investigate the autonomic and vascular function in men and women with Type 1 diabetes. The main questions it aims to answer are:

1. Patients with type 1 diabetes exhibit attenuated vascular function during steady-state exercise
2. Patients with type 1 diabetes have altered autonomic function at rest and during exercise pressor reflex
3. Patients with type 1 diabetes have attenuated muscle sympathetic activity

DETAILED DESCRIPTION:
Elevated blood glucose levels in individuals with type 1 diabetes can result in both microvascular and macrovascular complications. Research conducted by Song et al. revealed that children with type 1 diabetes exhibit abnormal cerebral perfusion. Additionally, autonomic mechanisms are affected in type 1 diabetes, as indicated in an animal study which demonstrated that the exercise pressor reflex is exaggerated in both male and female rats during the early stages of the disease. However, whether this also occurs in human patients with type 1 diabetes remains unknown.

Therefore, in this study we are interested in studying the autonomic control of exercise and vascular function in T1DM humans.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes or a Healthy control

Exclusion Criteria:

* BMI > 40kg/m2
* Cancer with current treatment
* HIV
* Smoker cigarettes
* Are pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 1 Diabetes
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular Function | Blood flow will be measured at baseline for 5 min in supine position. During exercise, blood flow will be measured continuously for the 3 minutes of handgrip exercise.
  Blood flow (ml/min) will be measured using Doppler ultrasound during steady-state dynamic exercise. Vascular conductance (ml/min/mmHg) will be calculated by dividing blood flow with blood pressure (mmHg). This measure will inform us about the vascular function in type 1 diabetic patients.
Autonomic Function | Blood presure will be measured at baseline for 10 minutes and continuously during 2 minutes of isometric handgrip.
  Blood pressure (mmHg) will be measured using Finapres at baseline and during activation of exercise pressor reflex. The exercise reflex will be activated by performing 2 minutes of isometric handgrip exercise at 30% and 40% of the maximal grip strength. This will inform us about the autonomic function in type 1 diabetic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided